CLINICAL TRIAL: NCT05692960
Title: Women's Interventions for Sexual Health: WISH, A Pilot Study
Brief Title: Women's Interventions for Sexual Health: WISH
Acronym: WISH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Tennessee, Knoxville (Other)
Collaborators: Breast Cancer Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UTK-IRB-22-07195
Record Dates: First submitted 2022-12-14; First posted 2023-01-20 (Actual); Results first posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-01

CONDITIONS: Sexual Dysfunction, Physiological; Body Image; Libido; Loss, Aversion
Keywords: breast cancer; vulvovaginal atrophy; libido; body image
MeSH Terms: conditions — Sexual Dysfunction, Physiological; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a two-arm, randomized clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Hypnotic Relaxation Intervention (HRI) (Experimental): The hypnotic relaxation intervention consists of three different audio files, each about 20 minutes in length. These three hypnotic inductions build upon each other. The first hypnotic induction audio focuses on relaxation, feelings of wellness, wholeness, strength, and confidence. The second hypnotic induction audio focuses more specifically on body image related to sexuality and being a sexual being. The third hypnotic induction audio focuses on sexual desire, passion, and energy. Each hypnotic induction will be used for two weeks, three times per week for a total of six weeks of hypnosis.
  The vaginal moisturizer component of this arm is the same as that described for the VVA study arm.
  Interventions: Other: Hypnotic Relaxation Intervention (HRI)
- Vulvovaginal Atrophy (VVA) (Other): This study arm might best be described as standard of care. Vulvovaginal dryness will be treated with a daily moisturizer for two weeks, then every other day for the remaining six weeks. Vaginal moisturizer will be applied at night, before sleep and after all sexual activity. Several moisturizers are available, including vaginal DHEA (IntraRosa®). Due to the need for reproducibility, we have decided to use one non-hormonal vaginal moisturizer, Replens™ moisture, which is a vaginal moisturizer consisting primarily of a purified water, glycerin, and mineral oil. Other ingredients included in the formulation are polycarbophyl, carbomer, homopolymer type B, hydrogenated palm oil glyceride, sorbic acid, sodium hydroxide. The moisturizing gel was determined to be a medical device for marketing by the FDA in 2010. It is non-hormonal (unlike vaginal DHEA) and therefore will be more likely to be acceptable by a broader range of oncology providers.
  Interventions: Device: Vulvovaginal Atrophy (VVA)

INTERVENTIONS:
Other: Hypnotic Relaxation Intervention (HRI) — HRI is a combination intervention (Replens™ vaginal moisturizer device and hypnotic relaxation behavioral intervention)
  Arms: Hypnotic Relaxation Intervention (HRI)
Device: Vulvovaginal Atrophy (VVA) — VVA is a standard of care intervention (Replens™ vaginal moisturizer device)
  Arms: Vulvovaginal Atrophy (VVA)

SUMMARY:
The overall objective of this program of research is to improve sexual health outcomes for women diagnosed with breast cancer. Our team is developing a multi-component intervention for the four key predictors of sexual health in female cancer survivors: self-image, vulvovaginal tissue quality and symptoms, desire/energy, and relationship-partner concerns. This proposal begins the proof-of-concept pilot study in women with a history of breast cancer to deliver a multi-component intervention to improve vulvo-vaginal atrophy with a vaginal moisturizer, and sexual energy and self-image with a mind-body intervention that involves relaxation and subconscious suggestions with a hypnotic induction delivered via audio file. The primary outcome will be to evaluate the feasibility and acceptability of a multi-component intervention for sexual function. It is hypothesized that at least eighty percent of randomized participants will complete the study without differential withdraws from the control group.

DETAILED DESCRIPTION:
Women's Interventions for Sexual Health (WISH), is a two-arm randomized clinical trial to evaluate the feasibility and acceptability of a multi-component intervention addressing changes in body image, sexual desire, and vaginal dryness in thirty adult post-treatment breast cancer survivors. The study is eight weeks long and does not require any in-person visits. If a breast cancer survivor is determined eligible, they will be educated on the purpose, requirements, and procedures. If interested, they will be emailed the consent form and will schedule a virtual consent/baseline visit. After consent is obtained, the participant will be randomly assigned to a study arm, HRI (hypnotic relaxation intervention plus vaginal moisturizer) or VVA (vulvovaginal atrophy moisturizer only), given a study number, and educated on the use of Replens™ vaginal moisturizer. The participant will complete online surveys at the virtual baseline visit. Replens™ vaginal moisturizer will be sent to the participant's address and receipt of the moisturizer will be confirmed by study staff before the agreed upon week one start date. The participant will use the moisturizer every day during weeks one and two and every other day during weeks three through eight. Participants randomized to the HRI group will also receive an MP3 player with three hypnotic relaxation audio files and asked to complete a weekly practice log. Each hypnotic induction audio file will be used for two weeks, three times per week, for a total of six weeks of hypnosis. A second virtual visit will be held at two weeks to assess progress, adverse events and provide education to the HRI group. Check in phone calls will be scheduled for weeks four, six and eight. A link to online follow up surveys will be shared during weeks six and eight.

ELIGIBILITY:
Inclusion Criteria:

* History of breast cancer, stages I, II or III
* Completed primary treatment (chemotherapy, radiation and/or surgery) ≥3 months and ≤ 5 years prior to registration
* May use concurrent adjuvant endocrine therapy or HER2-targeted therapy while on study
* May use topical products (e.g., lidocaine) vaginally prior to penetrative vaginal sex
* Ability to read and write English
* Able to engage in sexual activity
* Currently has a sexual partner Responds "yes" to "Do you currently experience vaginal or vulvar dryness and/or pain with sexual activity?"
* Responds "yes" to at least one of the following questions:

  1. "Have you experienced negative changes in your body image since being diagnosed or treated for cancer?" or
  2. "Have you experienced negative changes in your sexual desire since being diagnosed or treated for cancer?"

Exclusion Criteria:

* Antidepressants are allowed if a person has been on them for 30 days prior to registration, and dose or treatment is not expected to change
* History of sexual abuse
* Psychiatric disorder such as major depressive disorder, bipolar disorder, obsessive compulsive disorder or schizophrenia. (Defined per medical history and/or patient self-report)
* Currently enrolled in another study that addresses sexual health (enrollment in other clinical trials will be allowed)
* Use of oral, transdermal or vaginal estrogen is not allowed while on study

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2024-02-09 (Actual); Study Completion 2024-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Noel M Arring, DNP, PhD, RN, Principal Investigator — University of Tennessee Knoxville
Locations (1):
- University of Tennessee Knoxville, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
This is a small pilot study and as such, data will be thoroughly interrogated. However, if an investigator feels there are unanswered questions or wishes to add to a larger dataset, we would entertain all data sharing requests for deidentified data as appropriate.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through community recruitment efforts, social media, and ResearchMatch.org. The first participant was enrolled on February15, 2023 and the last on December 5, 2023.
Groups:
- Hypnotic Relaxation Intervention (HRI), Moisturizer and Self Hypnosis: The hypnotic relaxation intervention consists of three different audio files, each about 20 minutes in length. These three hypnotic inductions build upon each other. The first hypnotic induction audio focuses on relaxation, feelings of wellness, wholeness, strength, and confidence. The second hypnotic induction audio focuses more specifically on body image related to sexuality and being a sexual being. The third hypnotic induction audio focuses on sexual desire, passion, and energy. Each hypnotic induction will be used for two weeks, three times per week for a total of six weeks of hypnosis.
  The vaginal moisturizer component of this arm is the same as that described for the VVA study arm.
  Hypnotic Relaxation Intervention (HRI): HRI is a combination intervention (Replens™ vaginal moisturizer device and hypnotic relaxation behavioral intervention)
- Vulvovaginal Atrophy (VVA), Moisturizer Only: This study arm might best be described as standard of care. Vulvovaginal dryness will be treated with a daily moisturizer for two weeks, then every other day for the remaining six weeks. Vaginal moisturizer will be applied at night, before sleep and after all sexual activity. Several moisturizers are available, including vaginal DHEA (IntraRosa®). Due to the need for reproducibility, we have decided to use one non-hormonal vaginal moisturizer, Replens™ moisture, which is a vaginal moisturizer consisting primarily of a purified water, glycerin, and mineral oil. Other ingredients included in the formulation are polycarbophyl, carbomer, homopolymer type B, hydrogenated palm oil glyceride, sorbic acid, sodium hydroxide. The moisturizing gel was determined to be a medical device for marketing by the FDA in 2010. It is non-hormonal (unlike vaginal DHEA) and therefore will be more likely to be acceptable by a broader range of oncology providers.
  Vulvovaginal Atrophy (VVA): VVA is a standard of care intervention (Replens™ vaginal moisturizer device)
Period: Overall Study
Arm/Group | Hypnotic Relaxation Intervention (HRI), Moisturizer and Self Hypnosis | Vulvovaginal Atrophy (VVA), Moisturizer Only
Started | 14 | 16
Completed | 14 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hypnotic Relaxation Intervention (HRI), Moisturizer and Self Hypnosis | Vulvovaginal Atrophy (VVA), Moisturizer Only | Total
Number analyzed (Participants) | 14 | 16 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.79 (10.82) | 56.94 (10.83) | 55 (10.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 16 | 30
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 14 | 16 | 30
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 14 | 14 | 28
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 16 | 30
Sexual Orientation [Count of Participants; unit: Participants]
  Asexual | 0 | 0 | 0
  Bisexual | 0 | 1 | 1
  Fluid | 0 | 0 | 0
  Gay | 0 | 0 | 0
  Lesbian | 0 | 1 | 1
  Pansexual | 0 | 0 | 0
  Queer | 0 | 0 | 0
  Straight (heterosexual) | 14 | 14 | 28
  Prefer not to disclose | 0 | 0 | 0
  Other not listed | 0 | 0 | 0
Education Level [Count of Participants; unit: Participants]
  Did not complete high school | 0 | 0 | 0
  High school graduate or GED | 0 | 1 | 1
  Some college | 3 | 1 | 4
  Undergraduate degree | 5 | 4 | 9
  Master's degree | 6 | 9 | 15
  Doctorate | 0 | 1 | 1
  Prefer not to answer | 0 | 0 | 0
Marital status [Count of Participants; unit: Participants]
  Single, never married | 0 | 0 | 0
  Married | 14 | 15 | 29
  Divorced | 0 | 0 | 0
  Single, living with partner | 0 | 1 | 1
  Widowed | 0 | 0 | 0
  Other | 0 | 0 | 0
Cancer stage at time of diagnosis [Count of Participants; unit: Participants] — Participant stage based on the American Joint Committee on Cancer (AJCC) Tumor-Node-Metastasis system. Stage I: the tumor is small (2 cm or less) and hasn't spread to lymph nodes. Stage II: the tumor is larger (more than 2 cm) or has spread to nearby lymph nodes. Stage III: Locally advanced breast cancer, where the cancer has spread to nearby lymph nodes and potentially to the breast tissue or chest wall.
  Participants
    Stage I | 7 | 8 | 15
    Stage II | 6 | 7 | 13
    Stage III | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Screen Failure Rate (a Measure of Feasibility)
Description: The number of women screened ineligible / number of individuals for whom full eligibility criteria were evaluated
Time Frame: Up to 30 days Recruitment to screening
Measure: Count of Participants; unit: Participants
Groups:
- All Individuals Contacted: Across all recruitment methods, a total of 52 individuals participated in completing a screening checklist to determine their eligibility for the study. This number is not tied to study arm. Of these 52 individuals 36 were determined to be eligible.
Arm/Group | All Individuals Contacted
Number analyzed (Participants) | 52
Participants | 36

2. Primary Outcome: Accrual Rate (a Measure of Feasibility)
Description: The number of participants who consented divided by the number eligible
Time Frame: Up to 30 days Screening to consent
Measure: Count of Participants; unit: Participants
Arm/Group | All Individuals Contacted
Number analyzed (Participants) | 36
Participants | 30

3. Primary Outcome: Retention Rate/Acceptability (a Measure of Feasibility)
Description: The number of participants who completed the 8 weeks of the study divided by the number who consented.
Time Frame: Baseline through study completion, 8 weeks
Population: The number of participants who completed all 8 weeks of the study divided by the number who were randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Hypnotic Relaxation Intervention (HRI), Moisturizer and Self Hypnosis | Vulvovaginal Atrophy (VVA), Moisturizer Only
Number analyzed (Participants) | 14 | 16
Participants | 14 | 16

4. Secondary Outcome: Female Sexual Function Index (FSFI)
Description: The Female Sexual Function Index (FSFI) is a 19-item scale that measures the following domains of female sexual functioning: desire (subscale scale = 1.2-6), arousal (subscale = 0-6), satisfaction (subscale = 0.8-6), orgasm (subscale = 0-6), lubrication (subscale = 0-6) and pain (subscale = 0-6). When the scores of these domains are added together, the sum represents an FSFI total score.
  The following subscales were examined in this study: FSFI total (subscale range = 2-36 where higher scores indicate better sexual function); lubrication (subscale = 0-6 where higher scores indicate greater lubrication), pain (subscale = 0-6 where lower scores indicate greater pain); and desire (subscale scale = 1.2-6 where higher scores indicate greater desire).
Time Frame: consent to week 8
Population: All participants who were assigned to the study arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hypnotic Relaxation Intervention (HRI), Moisturizer and Self Hypnosis | Vulvovaginal Atrophy (VVA), Moisturizer Only
Number analyzed (Participants) | 14 | 16
score on a scale
  FSFI Total, Baseline | 14.56 (5.21) | 12.82 (6.97)
  FSFI Total, Week 8 | 22.35 (8.21) | 21.44 (7.34)
  FSFI Lubrication, Baseline | 2.06 (1.26) | 1.65 (1.33)
  FSFI Lubrication, Week 8 | 3.90 (1.71) | 3.92 (1.76)
  FSFI Pain, Baseline | 2.26 (1.58) | 1.80 (1.54)
  FSFI Pain, Week 8 | 3.54 (2.13) | 3.20 (2.23)
  FSFI Desire, Baseline | 2.06 (.84) | 2.03 (.95)
  FSFI Desire, Week 8 | 3.17 (1.09) | 3.08 (.75)
Statistical Analysis 1: Comparison: Hypnotic Relaxation Intervention (HRI), Moisturizer and Self Hypnosis; Effect sizes, Cohen's d, were calculated for both study arms using paired t-tests for FSFI total, FSFI lubrication, FSFI pain, and FSFI desire subscales. Means and 95% confidence intervals were also calculated; Test type: Superiority — For this feasibility study, a sample of approximately 15 participants per arm will allow for estimates that can be used in the development of a larger study; FSFI Total, HRI Cohen's d = 1.37, 95% CI 2-sided [.62 to 2.10]
Statistical Analysis 2: Comparison: Vulvovaginal Atrophy (VVA), Moisturizer Only; Test type: Superiority; FSFI Total, VVA Cohen's d = 1.63, 95% CI 2-sided [.86 to 2.37]
Statistical Analysis 3: Comparison: Hypnotic Relaxation Intervention (HRI), Moisturizer and Self Hypnosis; Test type: Superiority; FSFI Lubrication, HRI Cohen's d = 1.20, 95% CI 2-sided [.49 to 1.87]
Statistical Analysis 4: Comparison: Vulvovaginal Atrophy (VVA), Moisturizer Only; Test type: Superiority; FSFI Lubrication, VVA Cohen's d = 1.85, 95% CI 2-sided [1.02 to 2.66]
Statistical Analysis 5: Comparison: Hypnotic Relaxation Intervention (HRI), Moisturizer and Self Hypnosis; Test type: Superiority; FSFI Pain, HRI Cohen's d = .77, 95% CI 2-sided [.16 to 1.36]
Statistical Analysis 6: Comparison: Vulvovaginal Atrophy (VVA), Moisturizer Only; Test type: Superiority; FSFI Pain, VVA Cohen's d = .82, 95% CI 2-sided [.24 to 1.38]
Statistical Analysis 7: Comparison: Hypnotic Relaxation Intervention (HRI), Moisturizer and Self Hypnosis; Test type: Superiority; FSFI Desire, HRI Cohen's d = 1.15, 95% CI 2-sided [.46 to 1.82]
Statistical Analysis 8: Comparison: Vulvovaginal Atrophy (VVA), Moisturizer Only; Test type: Superiority; FSFI Desire, VVA Cohen's d = 1.21, 95% CI 2-sided [.55 to 1.86]

5. Secondary Outcome: Breast Impact of Treatment Scale (BITS)
Description: The Breast Impact of Treatment Scale (BITS) is a 13-item scale that measures body change stress in women with breast cancer. Scores range from 0-65. Higher scores indicate greater body change stress.
Time Frame: consent to week 8
Population: All participants who were assigned to the study arm.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hypnotic Relaxation Intervention (HRI), Moisturizer and Self Hypnosis | Vulvovaginal Atrophy (VVA), Moisturizer Only
Number analyzed (Participants) | 14 | 16
units on a scale
  BITS, Baseline | 30.71 (14.91) | 35.00 (16.54)
  BITS, Week 8 | 19.50 (14.85) | 28.81 (16.67)
Statistical Analysis 1: Comparison: Hypnotic Relaxation Intervention (HRI), Moisturizer and Self Hypnosis; Effect sizes, Cohen's d, were calculated for both study arms using paired t-tests for the BITS. Means and 95% confidence intervals were also calculated; Test type: Superiority — [test comment as in outcome 4, analysis 1]; BITS, HRI Cohen's d = 1.00, 95% CI 2-sided [.34 to 1.63]
Statistical Analysis 2: Comparison: Vulvovaginal Atrophy (VVA), Moisturizer Only; Test type: Superiority; BITS, VVA Cohen's d = .50, 95% CI 2-sided [.03 to 1.01]

6. Secondary Outcome: Patient Reported Outcomes Measurement Information System (PROMIS) Sexual Function and Satisfaction V2.0 (PROMIS SexF V2 )
Description: The PROMIS SexF V2 is a 14-item scale that includes screener items and measures sexual activities, symptoms, functioning, and evaluation of sexual experiences. It includes the following domains: interest in sexual activity, lubrication, vaginal discomfort, clitoral discomfort, labial discomfort, orgasm and pleasure, and satisfaction. Raw scores were converted to t-scores where the mean(standard deviation) = 50(10) in the referent population. Higher scores indicate more of the thing being described. Researchers are encouraged to select the sexual function and satisfaction domains and items that are relevant to the specific sample being studied. In this study, the interest, satisfaction and lubrication subscales were used.
Time Frame: consent to week 8
Population: All participants who were assigned to the study arm and completed PROMIS survey. The interest subscale was completed without missing data. Both the satisfaction and lubrication subscales begin with a screening question that asks "In the past 30 days, did you have any type of sexual activity?" A total of 5 participants responded "no" this item. For these subscales, total participants in HRI=13 and VVA=12.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hypnotic Relaxation Intervention (HRI), Moisturizer and Self Hypnosis | Vulvovaginal Atrophy (VVA), Moisturizer Only
Number analyzed (Participants) | 14 | 16
score on a scale
  PROMIS Interest Baseline | 31.33 (9.01) | 35.65 (7.51)
  PROMIS Interest Week 8 | 40.34 (11.10) | 41.48 (7.78)
  PROMIS Lubrication Baseline: number analyzed (Participants) | 13 | 12
  PROMIS Lubrication Baseline | 32.68 (7.11) | 34.28 (6.23)
  PROMIS Lubrication Week 8: number analyzed (Participants) | 13 | 12
  PROMIS Lubrication Week 8 | 45.65 (9.74) | 46.11 (8.63)
  PROMIS Satisfaction Baseline: number analyzed (Participants) | 13 | 12
  PROMIS Satisfaction Baseline | 38.23 (5.49) | 39.80 (4.19)
  PROMIS Satisfaction Week 8: number analyzed (Participants) | 13 | 12
  PROMIS Satisfaction Week 8 | 44.37 (8.14) | 47.16 (8.26)
Statistical Analysis 1: Comparison: Hypnotic Relaxation Intervention (HRI), Moisturizer and Self Hypnosis; Effect sizes, Cohen's d, were calculated for both study arms using paired t-test for PROMIS interest, lubrication and satisfaction subscales. Means and 95% confidence intervals were also calculated; Test type: Superiority — [test comment as in outcome 4, analysis 1]; PROMIS Interest, HRI Cohen's d = 1.10, 95% CI 2-sided [.41 to 1.75]
Statistical Analysis 2: Comparison: Vulvovaginal Atrophy (VVA), Moisturizer Only; Test type: Superiority; PROMIS Interest, VVA Cohen's d = .64, 95% CI 2-sided [.09 to 1.18]
Statistical Analysis 3: Comparison: Hypnotic Relaxation Intervention (HRI), Moisturizer and Self Hypnosis; Test type: Superiority; PROMIS Satisfaction, HRI Cohen's d = 1.19, 95% CI 2-sided [.45 to 1.89]
Statistical Analysis 4: Comparison: Vulvovaginal Atrophy (VVA), Moisturizer Only; Test type: Superiority; PROMIS Satisfaction, VVA Cohen's d = .80, 95% CI 2-sided [.13 to 1.44]
Statistical Analysis 5: Comparison: Hypnotic Relaxation Intervention (HRI), Moisturizer and Self Hypnosis; Test type: Superiority; PROMIS Lubrication, HRI Cohen's d = 1.79, 95% CI 2-sided [.88 to 2.67]
Statistical Analysis 6: Comparison: Vulvovaginal Atrophy (VVA), Moisturizer Only; Test type: Superiority; PROMIS Lubrication, VVA Cohen's d = 1.63, 95% CI 2-sided [.74 to 2.50]

ADVERSE EVENTS:
Time Frame: Adverse events were monitored every 2 weeks from week 1 to week 8.
Description: Adverse events were assessed during bi-weekly phone calls with participants and documented using the CTCAE version 5. All participants were assessed and included in the analysis.
Arm/Group | Hypnotic Relaxation Intervention (HRI), Moisturizer and Self Hypnosis | Vulvovaginal Atrophy (VVA), Moisturizer Only
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/16
Other Adverse Events (participants affected / at risk) | 8/14 | 7/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hypnotic Relaxation Intervention (HRI), Moisturizer and Self Hypnosis (N=14) | Vulvovaginal Atrophy (VVA), Moisturizer Only (N=16)
Anxiety (Psychiatric disorders) | 6 (7) | 3 (4)
Agitation (Psychiatric disorders) | 1 (1) | 3 (3)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 3 (5)
Sinusitus (Infections and infestations) | 0 (0) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-01-07): https://cdn.clinicaltrials.gov/large-docs/60/NCT05692960/Prot_SAP_000.pdf